CLINICAL TRIAL: NCT01420965
Title: A Pilot Study to Test the Feasibility and Immunologic Impact of Sipuleucel-T (Provenge) Administered With or Without Anti-PD-1 mAb (CT-011) and Low Dose Cyclophosphamide in Men With Advanced Castrate-Resistant Prostate Cancer
Brief Title: Sipuleucel-T, CT-011, and Cyclophosphamide for Advanced Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Samir N. Khleif, Cancer Center Director, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11C0231
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Prostatic Neoplasms
Keywords: Anti PD-1 Monoclonal Antibody; Vaccine; Autologous Cellular Immunotherapy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pidilizumab; spartalizumab; sipuleucel-T; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Sipuleucel-T autologous active cellular immunotherapy only for 3 cycles (cycle = 14 days)
  Interventions: Other: Sipuleucel-T (Provenge)
- Arm B (Experimental): Sipuleucel-T for 3 cycles (cycle = 14 days) + CT-011 (3mg/kg) IV infusion delivered over approximately 2 hours, 2 days after each Sipuleucel-T infusion
  Interventions: Drug: CT-011 (Anti-PD1 Antibody); Other: Sipuleucel-T (Provenge)
- Arm C (Experimental): Sipuleucel-T for 3 cycles (cycle = 14 days)+ cyclophosphamide (125 or 250mg/m2) IV [first cycle only] + CT-011 (3mg/kg) IV infusion delivered over approximately 2 hours, 2 days after each Sipuleucel-T infusion
  Interventions: Drug: CT-011 (Anti-PD1 Antibody); Other: Sipuleucel-T (Provenge); Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CT-011 (Anti-PD1 Antibody) — Immune Enhancer
  Other Names: Anti-PD1 Antibody
  Arms: Arm B; Arm C
Other: Sipuleucel-T (Provenge) — Vaccine
  Other Names: Provenge
Drug: Cyclophosphamide — Low dose- Immune Enhancer
  Other Names: Cytoxan
  Arms: Arm C

SUMMARY:
Background:

- Sipuleucel-T is a new treatment for advanced stage prostate cancer. It takes cells from a person with prostate cancer and treats them in the laboratory. Then it returns the cells to the person to help the immune system fight the cancer. Sipuleucel-T may be combined with the drug CT-011 to boost its ability to kill cancer cells. The chemotherapy drug cyclophosphamide will also be given, either before or after the cells are collected at the start of the treatment.

Objectives:

- To test the effectiveness of Sipuleucel-T, CT-011, and cyclophosphamide for prostate cancer.

Eligibility:

- Men at least 18 years of age who have advanced prostate cancer.

Design:

* Participants will be screened with a medical history, physical exam, blood and urine tests, and imaging studies.
* This study has two parts, with different participants in each part. All participants will be monitored with frequent blood tests and imaging studies.
* Part I:
* Participants will provide cells for the Sipuleucel-T treatment three times. The first time will be 3 days before the chemotherapy. The second time will be 10 days after chemotherapy. The third time will be 24 days after chemotherapy.
* Participants will have one dose of cyclophosphamide the day before the first dose of Sipuleucel-T.
* Participants will have Sipuleucel-T about 3 days after each cell donation.
* Part II:
* Participants will be in three groups: Sipuleucel-T given alone, given with CT-011, or given with both cyclophosphamide and CT-011.
* Participants will provide cells for the Sipuleucel-T treatment three times, as in Part I.
* Participants will have Sipuleucel-T about 3 days after each cell donation, and will receive treatment with the other drugs as directed by the study doctors.

DETAILED DESCRIPTION:
Background:

* Prostate cancer is the most common cancer and the second leading cause of cancer deaths among males in most Western countries.
* Sipuleucel-T, a recently FDA approved treatment for prostate cancer, is designed to induce an immune response targeted against PAP, an antigen expressed in most prostate cancers. .
* Blockade of PD-1/PD-L1 has been shown to enhance the therapeutic efficacy of peptide cancer vaccines in pre-clinical animal models. CT-011 is a humanized IgG1 kappa recombinant monoclonal antibody against PD-1 receptor that blocks the interaction of PD-L1 with PD-1.
* Preclinical studies demonstrated that CT-011 when administered with low dose cyclophosphamide led to synergistic antitumor effects when combined with HPV16 E749-57 peptide vaccine.
* Given the role CT-011 plays in down-regulating peripheral tolerance and the synergistic relationship it has with cyclophosphamide in doing so, in this study we propose to treat patients with advanced, castrate-resistant disease with CT-011 and low-dose cyclophosphamide as adjuvants in combination with Provenge(Trademark) activated cell vaccine.

Objectives:

* To assess the feasibility of administration of Sipuleucel-T (Provenge(Trademark)) autologous active cellular immunotherapy in combination with low dose cyclophosphamide in men with advanced castrate-resistant (hormone refractory) prostate cancer.
* To determine the immune efficacy of Sipuleucel-T (Provenge(Trademark)) autologous active cellular immunotherapy alone vs. Sipuleucel-T (Provenge(Trademark)) in combination with CT- 011 vs. Sipuleucel-T (Provenge(Trademark)) in combination with low-dose cyclophosphamide and CT-011 on the change in PA2024-specific IFN-? ELISPOT responses in men with advanced, castrate-resistant prostate cancer.
* Secondary objectives will determine the tolerability and toxicities of the combination of low-dose cyclophosphamide/CT-011/ Sipuleucel-T (Provenge(Trademark)) and determine in a preliminary fashion whether this regimen correlates with increased progression-free survival (PFS) and overall survival (OS) in patients and with growth rate in an exploratory fashion.

Eligibility:

* Males greater than or equal to 18 years old with chemotherapy na ve metastatic progressive castrate-resistant prostate cancer defined as progressive disease (two consecutively rising PSA values at a minimum of 1-week intervals (2.0 ng/mL is the minimum starting value for PSA), appearance of one or more new lesions on bone scans, progressive disease by Recist 1.1).
* Must meet minimum organ safety requirements and length of time since prior therapy.
* May not have active infections, autoimmune disease or require immunosuppressive therapies.

Design:

Part 1: Initially the feasibility generating Sipuleucel-T after administration of low dose cyclophosphamide , and will be evaluated using a standard 3 + 3 design for doses of cyclophosphamide 250 mg/m2 or 125 mg/m2. Initially 3 patients will receive cyclophosphamide on day -1 of the first cycle (one day prior to the first infusion of Sipuleucel-T). All patients will receive Sipuleucel-T cell infusion on Day 0. The Sipuleucel-T cell infusion will be repeated every two weeks for a total of three cycles. If Sipuleucel-T active cellular immunotherapy from an apheresis obtained after infusion of cyclophosphamide, which meets the FDA approved Certificate of Analysis (COA) release criteria from Dendreon, cannot be generated, a second apheresis will be performed. Failure of two attempts to generate Sipuleucel-T product after two aphereses at either the 2nd or 3rd scheduled Sipuleucel-T infusion will be considered failure of one patient to meet release criteria .

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histopathological documentation of prostate cancer prior to starting this study.

Patients must have metastatic progressive castrate-resistant prostate cancer defined as progressive disease (see below) despite surgical castration or ongoing use of gonadotropin-releasing hormone agonists with confirmed castrate levels of testosterone. Criteria of progression for trial eligibility are defined from the Prostate Cancer Clinical Trials Working Group-253. Clinically progressive prostate cancer must be evidenced and documented by any of the following parameters:

1. Two consecutively rising PSA values at a minimum of 1-week intervals (2.0 ng/mL is the minimum starting value for PSA)
2. Appearance of one or more new lesions on bone scans
3. Progressive measurable disease by RECIST 1.1

   Patients on flutamide for at least 6 months must have disease progression at least 4 weeks after withdrawal. Patients on bicalutamide or nilutamide for at least 6 months must have progression at least 6 weeks after withdrawal.2.1.1.4 Performance Status: ECOG 0-1 or Karnofsky 80-100% (asymptomatic or minimally symptomatic from metastatic disease).

   No previous chemotherapy use.

   No therapeutic immunosuppression or immunomodulation altering bone marrow function within 6 weeks prior to study entry e.g. G-CSF, GM-CSF, EPO, prednisone etc.

   Must have adequate:
   * Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl. Platelets greater than or equal to 100,000/mcl.
   * Renal function: Creatinine less than or equal to 1.5 times institutional upper limit normal (ULN)
   * Hepatic function: Bilirubin less than or equal to 1.5 x ULN (CTCAE v4.0 grade 1) except patients with Gilbert's disease (up to 5.0 mg/dL). SGOT and alkaline phosphatase less than or equal to 2.5 x ULN.
   * Normal Cardiac function: ECG with no evidence of arrhythmia, conduction abnormality or ischemia. No active coronary artery disease; no New York Heart Association class II, III or IV disease; no arrhythmia requiring treatment.

   Must willing and able to sign an informed consent document that explains the neoplastic nature of the disease, the procedures to be followed, the experimental nature of the treatment, alternative treatment and potential risks and toxicities.

   EXCLUSION CRITERIA:

   Concurrent treatment with any other cancer therapies including radiation (except palliative radiation therapy for bone metastases), chemotherapy or other investigational agent(s). Androgen suppression therapy will be allowed.

   History of a second active malignancy in the last 2 years other than non-melanoma skin cancers.

   Patients who have active or history of autoimmune disease/symptom/conditions including: type I diabetes, rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis. Type II diabetes mellitus, vitiligo or stable hypothyroidism are not considered exclusion criteria.

   Patients being chronically treated with immunosuppressive drugs such as cyclosporin, adrenocorticotropic hormone (ACTH).

   Concurrent use of systemic glucocorticoids within 4 weeks prior to trial entry

   Patients who have acquired, hereditary, or congenital immunodeficiencies including cellular immunodeficiencies, hypogammaglobulinemia and dysgammaglobulinemia.

   CNS, lung, or liver metastasis, because of the poor prognosis, and potential inability to meet study endpoints.

   Serious active infection at the time of pre-study screening.

   Positive HIV or Hepatitis C antibodies or Hepatitis B anti-core antibodies, because immunotherapies rely on intact immune systems, and toxicities may be exacerbated by the presence of infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir N. Khleif, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Center MM, DeSantis C, Ward EM. Global patterns of cancer incidence and mortality rates and trends. Cancer Epidemiol Biomarkers Prev. 2010 Aug;19(8):1893-907. doi: 10.1158/1055-9965.EPI-10-0437. Epub 2010 Jul 20. PMID 20647400
- [Background] Gittes RF. Carcinoma of the prostate. N Engl J Med. 1991 Jan 24;324(4):236-45. doi: 10.1056/NEJM199101243240406. No abstract available. PMID 1985245
- [Background] Crawford ED, Eisenberger MA, McLeod DG, Spaulding JT, Benson R, Dorr FA, Blumenstein BA, Davis MA, Goodman PJ. A controlled trial of leuprolide with and without flutamide in prostatic carcinoma. N Engl J Med. 1989 Aug 17;321(7):419-24. doi: 10.1056/NEJM198908173210702. PMID 2503724

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 2 | 2 | 3
Completed | 1 | 1 | 3
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 2 | 2 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 5
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 2 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 1 | 3 | 5
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Determine Feasibility of Provenge Plus Low-dose Cyclophosphamide as Well as the Immune Efficacy of Provenge Alone Versus Provenge Plus Low-dose Cyclophosphamide and Anti PD1 Monoclonal Antibodies (CT011) on the Change in Specific Immune Response.
Time Frame: 2 years
Population: Study discontinued due to drug supply issues; no analysis performed or meaningful data derived.
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Determine Whether the Combination of Low Dose-Cyclophosphamide and Anti PD1 Monoclonal Antibodies (CT-011) With Provenge(tm) Lead to Improvement in Increase Progression Free Survival (PFS) and Overall Survival (OS) in Patients With Advanced, Min...
Time Frame: 2 years
Population: Study discontinued due to drug supply issues; no analysis performed or meaningful data derived.
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B | Arm C
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=2) | Arm B (N=2) | Arm C (N=3)
Negative infusion reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other